# **STUDY TITLE:**

PREVENTION OF DEPRESSION AND BULLYING IN ADOLESCENTS BY MEANS OF AN INTERVENTION BASED ON IMPLICIT THEORIES OF PERSONALITY

## **PROJECT NUMBER:**

PSI2015-68426-R

(Ministry of the Economy and Competitiveness, Spanish Government)

## PI:

Esther Calvete Zumalde, PhD, University of Deusto Research team:

Izaskun Orue Sola, PhD, University of Deusto Liria Fernández-González, PhD, University of Deusto Anik Zubizarreta Arturo, MD, PhD, University of Deusto

## **Collaborators:**

David Scott Yeager, PhD, University of Texas at Austin
Todd Little, PhD, Texas Tech University

SEPTEMBER, 2016

#### I. BACKGROUND

Depression and aggressive behavior are psychological problems of crucial clinical and social relevance. According to data from the World Health Organization (WHO, 2012), more than 350 million people suffer from major depressive disorder, which constitutes one of the most important causes of disability. Depression involves great suffering in people, contributing to significant difficulties in their social, academic, and professional life. There is a dramatic increase of depression rates in adolescence. Moreover, depression in adolescence is the most powerful predictor of experiencing depression in adulthood. On the other hand, aggressive behavior is also highly prevalent in our society. Often arises early but increases in severity over time. As children enter adolescence aggressions towards peers give way to other modalities such as dating violence and violence against parents. Therefore, preventing the development of depression and aggressive behavior in childhood and adolescence is invaluable. Unfortunately, although there are adequate interventions for adolescents at risk of depression, results for the majority of the previous universal interventions have been poor. In the case of aggressive behavior current preventive interventions are expensive in terms of duration and involve working with children, their parents, and educators.

The current project will test the efficacy of an Implicit Theory of Personality (ITP) intervention, which has provided excellent results in US both for depression and externalizing problems such as aggressive behavior. The project includes two studies, one focused on depression and another one focused on aggressive behavior. In addition, we will evaluate at which developmental stage the intervention is more effective. Finally, we will examine the moderation role of sex. The project includes biological data in a subsample of participants. Therefore, the project will contribute from a biopsychosocial and interdisciplinary perspective to the development of universal preventive interventions for depression and aggressive behavior, two important psychological problems in modern societies.

## Preventive approaches to depression and aggressive behavior

Several depression prevention programs have been developed, such as the Coping with Stress program (Clarke et al., 1995), the Blues Program (Stice, Burton, Bearman, & Rohde, 2007), the UK Resilience Program (Challen, Machin, & Gillham, 2014), and the Penn Resiliency Program (Cardemil, Reivich, Beevers, Seligman, & James, 2006). Most prevention programs have targeted factors that have been found to increase risk for future onset of depression or increases in depressive symptoms, such as negative cognitions, social skill deficits, and ruminative style. The results from meta-analytic reviews of the effects of depression prevention programs for youth indicate that although results are good for indicated and selective preventive interventions, the average effects of universal preventive interventions on depressive symptoms from pretest to posttest are small (Mychailyszyn, Brodman, Read, &

Kendall, 2012; Stice, Shaw, Bohon, Marti, & Rohde, 2009). Interestingly, Stice et al. (2009) found that relatively shorter prevention programs produced significantly larger intervention effects than did longer prevention programs. Therefore, the authors concluded that long programs may not appeal to youth, which causes greater attrition and attenuated intervention effects. Thus, they recommended the use of brief interventions for future studies.

Regarding aggressive behavior several multicomponent interventions with elements directed towards children and adolescents as well as towards their parents and teachers have been developed and have been found to be effective. Some noteworthy examples are the Coping Power (Lochman & Wells, 2002), the Fast Track (Conduct Problems Prevention Research Group, 2002), the Montreal Preventive Treatment Program (Tremblay, Masse, Pagani, & Vitaro, 1996) and the Incredible Years programs (Webster-Stratton, Reid, & Stoolmiller, 2008). Although these programs have demonstrated to be useful, they are expensive in terms of duration and involvement of various actors (parents, schools, students).

## **Need of universal brief interventions**

In recent years numerous short-term psychosocial interventions have been developed in educational settings with striking effects on several outcomes such as student performance, social integration, and psychological wellbeing (see for a revision Yeager & Walton, 2011). Rigorous field experiments have shown that the effects of such interventions persist for months or even years later. For example, Blackwell, Trzesniewski, and Dweek (2007) got to substantially improve school skills through an intervention based on implicit theories of intelligence, which consisted of showing that intelligence is modifiable and grows when the individual works with effort in challenging tasks. In another intervention, Walton and Cohen (2007, 2011) found that leading students to attribute worries about social integration to the difficulty of the transition to college rather than to students' personal or racial identity can strengthen ethnic minority students' sense of social belonging in school and increase motivation and performance. Furthermore, students who received the intervention reported being happier and healthier in a 3 years posttreatment follow up.

These psychosocial interventions in school can be brief yet impactful because they rely on a rich tradition of research on persuasion and attitude change to powerfully convey psychological ideas (Yeager & Walton, 2011). The crucial elements that contribute to the success of these interventions are the focus on students' experience in school from the students' perspective and the use of impactful delivery mechanisms (Yeager & Walton, 2011). Some of these mechanisms are the following: a) Active role of students, which facilitates deeper message processing; b) Interventions are stealthy. For example, interventions are not presented to the students with the intent to improve performance or other attributes. Thus, students do not feel they are being manipulated so that resistance to intervention is reduced. This approach

contributes also to avoid the stigmatization of students. Moreover, the brevity of the interventions also helps to be stealthy. c) Psychosocial interventions have effects over long periods due to recursive processes affecting effects that accumulate over time. Students usually forget the message and the details of the intervention, but this recursive nature triggers other social, psychological and cognitive mechanisms over time.

# Implicit theory of personality (ITP) interventions for emotional and behavioral problems

Recently, Yeager and colleagues have extended this type of brief interventions to prevent emotional and behavioral problems such as depression and aggressive behavior in adolescents. Their approach is based on implicit theories of personality, which refer to the beliefs that people endorse about the malleability of people's socially-relevant traits. An entity theory of personality involves the belief that personal characteristics are fixed and cannot be changed whereas an incremental theory of personality involves the belief that people can change. Past research has found that when adolescents or adults believe that people's traits are fixed and unchangeable, they are more likely to attribute a negative social event (e.g., peer victimization) to their negative traits. They also will tend to infer that the same negative events and other adversities will repeat in the future. Therefore, an entity theory of personality predicts greater shame and negative emotions in adolescents when they cope with stressors such as peer conflicts (Yeager, Trzesniewski, Tirri, Nokelainen, & Dweck, 2011). By the contrary, if adolescents believe that traits can be changed, then their own traits can be improved so that it is unlikely that they become recipients of the same negative events in the future. Furthermore, other people' traits, including those of bullies, can also change. Therefore, the beliefs involved in an incremental theory of personality can be helpful not only for victims but also for perpetrators of bullying. As additional support to this, Rudolph (2010) found that holding an entity theory of peer relationships was associated with a greater tendency to evaluate oneself negatively in the face of peer disapproval and display depressive and aggressive symptoms when victimized.

Yeager and colleagues have developed brief interventions aimed to change entity theories by means of efficient and persuasive intervention tactics that are based on the above mentioned mechanisms. For instance, in one of these interventions, a six-session high school classroom intervention teaching an incremental theory reduced aggressive behavior by 40%, improved depressive symptoms two weeks post-intervention, and increased school attendance (Yeager, Trzesniewski, & Dweck, 2013). Later, they tested the effects of a shorter intervention consisting of only one session. This single session touch an incremental theory via computers. In this session 9<sup>th</sup> grade students read a scientific article about the possibility of personality change, then they read quotes from older students transmitting the same message. Finally, the students

wrote a brief essay where they defended the same idea with the aim of transmitting the message to other students in the future. Despite the brevity of this intervention, the results obtained by means of a double-blind randomized experiment showed that it reduced levels of self-reported clinically relevant depression (Miu & Yeager, 2014) and stress levels (Yeager et al., 2014).

#### **II. AIMS AND HYPOTHESES**

Aim 1: To replicate the effect of an intervention based on Implicit Theories of Personality (ITP) on depressive symptoms (Study 1) and aggressive behavior (Study 2) in a large sample of Spanish adolescents. Grounded on the previous findings obtained in US samples, we will test the efficacy of the ITP intervention by comparing changes in depressive symptoms and aggressive behavior from pretreatment to follow up between the group receiving the ITP intervention and a control group that will receive a control educational condition.

Hypothesis: Those adolescents receiving the ITP intervention will show fewer symptoms of depression and lower frequency of aggressive behavior than the control group after the intervention and at six-month and one-year follow-up.

Aim 2: To test whether the intervention changes biological and cognitive variables. From a biopsychosocial perspective, several mechanisms can explain the effect of the ITP intervention on psychological problems (depression and aggressive behavior). These mechanisms include changes in cognitive vulnerabilities and changes in the biological responses to the environmental stressors. If participants develop beliefs that personality traits are malleable, this should influence many maladaptive cognitive schemas. In fact, a feature of most maladaptive cognitive schemas is their absolute and stable nature (e.g., "I am a bad person", "The others will always reject me", "People hurt me on purpose", "I cannot put limits to my conduct". The intervention could also change biological indicators of stress (e.g., hormonal indicators). Therefore, in this project we will evaluate whether the ITP intervention affects cognitive vulnerabilities and biological indicators (cortisol, testosterone and DHEA in saliva).

Hypothesis: the association between the intervention and changes in psychological problems will be associated with changes in cognitive and hormonal variables. Some studies have explored whether the effects of interventions on depressive symptoms are mediated by changes in cognitive vulnerabilities with mixed results (Mychailyszyn et al., 2012). Thus, this project aims to contribute to clarifying mediational cognitive mechanisms.

**Aim 3:** To identify whether development and sex moderates the effects of the intervention. Regarding the developmental stage at which the preventive intervention is more effective, though studies are inconclusive, in general there is some consensus that cognitive vulnerabilities tend to consolidate in adolescence. Also in the case of

depression prevalence rates increase dramatically during adolescence. This supports the tentative hypothesis that the preventive intervention may be more effective if implemented early (i.e., before depression rates increase and cognitive vulnerabilities are consolidated).

As girls display higher rates of depression and boys higher rates of some modalities of aggressive behavior, sex could moderate the effects of the ITP intervention on psychological problems. For instance, we hypothesize that the ITP intervention will lead to a higher reduction of depressive symptoms in girls.

**Aim 4:** To test whether temperament moderates the effect of the intervention. We hypothesize that the intervention will be more effective in adolescents high in neuroticism.

#### III. METHODS

This project will use a randomized controlled trial study design with pretest, posttest, six-month follow-up, and one-year follow-up. Group 1 (experimental group) will receive the ITP intervention and Group 2 (control group) will receive an educational intervention.

### Study design and participants

We will conduct a double-blind randomized controlled trial (RCT) with two parallel groups in a large sample of volunteer adolescents (approximately n=900), from several high school centers (ages from 12 to 18 years). The schools will be randomly selected from the Basque Country. Participants will be randomly assigned to the experimental vs control groups. Group assignation will be done at the individual level within each classroom. Participants were randomized in a 1:1 ratio blocked by gender to one of two groups (experimental versus control condition). They were assigned to their allocated group in class by the researchers.

## Measures

Depressive symptoms and aggressive behavior will be assessed by means of self-reports through the Center for Epidemiologic Studies Depression scale (CES-D; Radloff, 1977), the revised version of the Peer Experiences Questionnaire (RPEQ; Prinstein, Boergers, & Vernberg, 2001), the Cyber Bullying Questionnaire (CBQ; Calvete, Orue, Estévez, Villardón, & Padilla, 2010; Gámez-Guadix, Villa-George, & Calvete, 2014.

Measures of cortisol, DHEA and testosterone in saliva: A subset of the participants (around 50%) will provide saliva samples to be assayed for neuroendocrine levels to measure cortisol, DHEA and testosterone. Saliva samples will be collected at baseline (one week before the intervention), post-intervention (one week after the intervention) and at the two follow-ups (six-months and one-year follow-up). Data collection will occur in school and the time of assessments will remain

the same for each individual to minimize the effects of diurnal rhythms and reduce error variance. The adolescents will complete an intake survey (e.g., eating, drinking, exercise, and medication) that can potentially affect hormonal reactivity. The adolescents will then be directed to transfer saliva from their mouths to a tube. The sample tubes will be carefully labelled. As soon as the session ends, saliva samples will be sent to the assay laboratory.

**Cognitive vulnerabilities**: Two important cognitive vulnerabilities will be assessed: dysfunctional cognitive schemas and beliefs about implicit theories of personality. We will measure cognitive schemas that are relevant for depression (i.e., defectiveness, emotional privation) in the study about depression. We will use the Spanish version of the Young Schema Questionnaire (YSQ; Young, 2006). In addition, we will measure implicit theories of personality through the Implicit Theories of Personality questionnaire (Yeager et al., 2014).

**Temperament traits:** Temperament will be assessed by the revised version of the Early Adolescent Temperament Questionnaire (EATQ-R; Ellis & Rothbart, 2001) and the Big Five Questionnaire for children (BFQ-C; Barbaranelli, Caprara, Rabasca, & Pastorelli, 2003) for adolescents at the beginning of the study.

Parent reports: Parents will be invited to participate by responding measures about their children temperament by means of the revised version of the Early Adolescent Temperament Questionnaire (EATQ-R; Ellis & Rothbart, 2001) and the Big Five Questionnaire for children (BFQ-C; Barbaranelli et al., 2003) for parents and depressive symptoms through the CBCL 6/18 (Achenbach, 1991; Achenbach & Edelbrock, 1983). These data will be used in analyses in case that the response rate is enough.

#### **Preventive Intervention**

The ITP intervention lasts one session (of approximately one hour) and has three main parts: (1) scientific information; (2) normative stories from upperclassmen; and (3) self-persuasive writing exercise. In the first part, students read a scientific article that provides evidence that individuals have the potential to change. Participants read about actual neurological and behavioral studies showing that behaviors are controlled by "thoughts and feelings in brains," and that pathways in the brain have the potential to be changed under the right circumstances. In the second part, participants read several normative quotes purportedly written by upperclassmen that previously read the same article and endorsed its conclusions. These quotes are obtained from previous interventions and edited by the team. These testimonials are provided to bring credibility to the incremental theory. Finally, in the last part, participants will be asked to write their own version of such a narrative to share with future students, This activity has been shown to facilitate the internalization of the intervention message,

building on a long line of research on cognitive dissonance (Walton & Cohen, 2011). For a more complete description of the ITP intervention see Yeager et al. (2013). The intervention will be adapted to the developmental characteristics of the participants.

The **educational intervention** involves scientific information about the human brain. It was designed to be parallel to the experimental intervention and, hence, it has also three main parts. First, participants are asked to read scientific information about the different areas of the brain and their specialties. Second, participants read several testimonials written by upperclassmen about their transition to high school and how their brains help them to adapt to the new space and all the physical differences of the building and the classes. Finally, participants are asked to write a letter to another student explaining the main things he or she has learned about the brain and thinks are important for adapting to the new physical environment in high school. Hence it will control for the possibility that simple optimism about the potential for growth might account for our results. This is a conservative control group. An entity theory control group would be unethical in a longitudinal field experiment because it could teach the belief that personality cannot be changed, which has been associated to negative consequences.

#### **Procedure**

Parental informed consent forms will be sent to parents and adolescents. Those who accept to participate in the study will complete report measures at four waves: (1) one-week before intervention; (2) one-week after intervention; (3) six-months follow-up; and (3) one-year follow-up. Saliva samples will be collected at the same time points. Parents' participants will complete report measures at three waves: (1) one-week before intervention; (2) six-months follow-up; and (3) one-year follow-up. Intervention will be applied one week after the first survey. All the measures will be anonymous and participants will be asked to provide certain data (her/his birth date, first initial of mother's name, and first initial of father's name) to match their questionnaires, saliva samples and intervention tasks over time. Both interventions and assessment measures will be administered by research assistants during normal class time and last around 50 minutes.

## **Ethical considerations**

This study aims to develop and implement interventions that will be beneficial for the participating adolescents and other people in the future, by helping to increase their psychological wellbeing. Through randomization, the principle of justice will be respected, allowing all participants to have similar opportunities to receive the intervention. Gender will be considered and similar number of male and female participants will be included in the studies.

The risks are minimal and limited to answering psychological tests on stressors, psychological symptoms and cognitive styles. Previous experience with the same

questionnaires indicates that the risk is minimal. Adolescents can also decide to end their participation at any moment. Researchers collecting data will be trained to attend to any difficulty that could emerge while participants are responding to questionnaires. The researchers will give an alternative task (e.g., educational readings) to those participants who decide to end their participation.

Informed consent forms will be sent to parents or legal guardians to complete. Adolescents will also receive written information. The active consent of parents or legal guardians and of adolescents will be necessary for participation in the project. We will incentive adolescents for bringing parent forms, even when decision is negative.

Parents will be invited to complete measures of children'temperament and send their completed questionnaires in a stamped envelope that will be provided without any identifying information. Adolescents will complete the measures in the classroom. Saliva samples and their analysis will be processed according to existing regulations in a professional lab.

After completing measures, adolescents will be provided with information on services for adolescents (e.g., phone number of attention to adolescents). From an ethical perspective, the most important care aspect is the protection of information. We will follow the Directive 95/46/EC of the European Parliament, *Ley Orgánica 15/99 de 13 de diciembre de Protección de datos de Carácter Personal*, and of the Council of 24 October 1995 on the protection of individuals with regard to the processing of personal data and the free movement of such data. No identification data, such as names or surnames, will be used; instead, we will use a numeric code to match measures across times and sources (parents, and adolescents). Thus, each adolescent, and only he/she, will know his/her code. We will also follow the procedure for data protection that the University of Deusto has registered in the National Data Protection Agency. The project has been approved by the Ethics in Research committee of University of Deusto.

## IV. STATISTICAL ANALYSES PLAN

Descriptive statistics of sociodemographic and study variables will be provided and several statistical strategies will be used to test the hypotheses. These will include mixed analyses of variance (ANOVA), multilevel analyses, regression analyses, among others. We will use IBM SPSS, MPLUS, LISREL, and HLM software for analyses.

#### References

- Achenbach, T. M. (1991). Child Behavior Checklist/4-18 and 1991 profile. *Burlington, Vermont, USA: University of Vermont, Department of Psychiatry*.
- Achenbach, T. M., & Edelbrock, C. S. (1983). Manual for the Child Behavior Checklist/4-18 and revised child behavior profile. *Burlington, Vermont, USA: University of Vermont, Department of Psychiatry*.
- Barbaranelli, C., Caprara, G. V., Rabasca, A., & Pastorelli, C. (2003). A questionnaire for measuring the Big Five in late childhood. *Personality and Individual Differences,* 34(4), 645-664. doi:10.1016/s0191-8869(02)00051-x
- Blackwell, L. S., Trzesniewski, K. H., & Dweck, C. S. (2007). Implicit theories of intelligence predict achievement across an adolescent transition: A longitudinal study and an intervention. *Child Development*, *78*(1), 246-263. doi:10.1111/j.1467-8624.2007.00995.x
- Calvete, E., Orue, I., Estévez, A., Villardón, L., & Padilla, P. (2010). Cyberbullying in adolescents: Modalities and aggressors' profile. *Computers in Human Behavior*, 26(5), 1128-1135. doi:10.1016/j.chb.2010.03.017
- Cardemil, E. V., Reivich, K. J., Beevers, C. G., Seligman, M. E., & James, J. (2006). The prevention of depressive symptoms in low-income, minority children: Two-year follow-up. *Behaviour Research and Therapy*, *45*(2), 313-327. doi:10.1016/j.brat.2006.03.010
- Challen, A. R., Machin, S. J., & Gillham, J. E. (2014). The UK Resilience Programme: A school-based universal nonrandomized pragmatic controlled trial. *Journal of Consulting and Clinical Psychology*, 82(1), 75-89. doi:10.1037/a0034854
- Clarke, G. N., Hawkins, W., Murphy, M., Sheeber, L. B., Lewinsohn, P. M., & Seeley, J. R. (1995). Targeted prevention of unipolar depressive disorder in an at-risk sample of high school adolescents: A randomized trial of a group cognitive intervention. *Journal of the American Academy of Child and Adolescent Psychiatry, 34*(3), 312-321. doi:10.1097/00004583-199503000-00016
- Conduct Problems Prevention Research Group. (2002). Using the Fast Track randomized prevention trial to test the early-starter model of the development of serious conduct problems. *Development and Psychopathology*, *14*(4), 925-943. doi:10.1017/s0954579402004133
- Ellis, L. K., & Rothbart, M. K. (2001). Revision of the Early Adolescent Temperament Questionnaire. *Biennial Meeting of the Society for Research in Child Development* (2001). Minneapolis, Minnesota, USA.
- Gámez-Guadix, M., Villa-George, F., & Calvete, E. (2014). Psychometric properties of the Cyberbullying Questionnaire (CBQ) among Mexican adolescents. *Violence and Victims*, *29*(2), 232-247. doi:10.1891/0886-6708.vv-d-12-00163r1
- Lochman, J. E., & Wells, K. C. (2002). The Coping Power program at the middle-school transition: Universal and indicated prevention effects. *Psychology of Addictive Behaviors*, *16*(4S), S40-S54. doi:10.1037/0893-164x.16.4s.s40

- Miu, A., & Yeager, D. S. (2014). Preventing symptoms of depression by teaching adolescents that people can change: Effects of a brief incremental theory of personality intervention at 9-month follow-up. *Clinical Psychological Science*, 3(5), 726-743. doi:10.1177/2167702614548317
- Mychailyszyn, M. P., Brodman, D. M., Read, K. L., & Kendall, P. C. (2012). Cognitive-behavioral school-based interventions for anxious and depressed youth: A meta-analysis of outcomes. *Clinical Psychology: Science and Practice*, 19(2), 129-153. doi:10.1111/j.1468-2850.2012.01279.x
- Prinstein, M. J., Boergers, J., & Vernberg, E. M. (2001). Overt and relational aggression in adolescents: Social-psychological adjustment of aggressors and victims. *Journal of Clinical Child Psychology, 30*(4), 479-491. doi:10.1207/s15374424jccp3004 05
- Radloff, L. S. (1977). The CES-D Scale: A self-report depression scale for research in the general population. *Applied Psychological Measurement*, *1*(3), 385-401. doi:10.1177/014662167700100306
- Rudolph, K. D. (2010). Implicit theories of peer relationships. *Social Development*, *19*(1), 113-129. doi:10.1111/j.1467-9507.2008.00534.x
- Stice, E., Burton, E., Bearman, S. K., & Rohde, P. (2007). Randomized trial of a brief depression prevention program: An elusive search for a psychosocial placebo control condition. *Behaviour Research and Therapy, 45*(5), 863-876. doi:10.1016/j.brat.2006.08.008
- Stice, E., Shaw, H., Bohon, C., Marti, C. N., & Rohde, P. (2009). A meta-analytic review of depression prevention programs for children and adolescents: Factors that predict magnitude of intervention effects. *Journal of Consulting and Clinical Psychology*, 77(3), 486-503. doi:10.1037/a0015168
- Tremblay, R. E., Masse, L., Pagani, L., & Vitaro, F. (1996). From childhood physical aggression to adolescent maladjustment: The Montreal Prevention Experiment. In R. D. Peters & R. J. McMahon. (Eds.), *Preventing childhood disorders, substance abuse, and delinquency* (pp. 268-298). Thousand Oaks, California, USA: Sage Publications.
- Walton, G. M., & Cohen, G. L. (2007). A question of belonging: Race, social fit, and achievement. *Journal of Personality and Social Psychology*, *92*(1), 82-96. doi:10.1037/0022-3514.92.1.82
- Walton, G. M., & Cohen, G. L. (2011). A brief social-belonging intervention improves academic and health outcomes of minority students. *Science*, *331*(6023), 1447-1451. doi:10.1126/science.1198364
- Webster-Stratton, C., Reid, J., & Stoolmiller, M. (2008). Preventing conduct problems and improving school readiness: Evaluation of the Incredible Years Teacher and Child Training Programs in high-risk schools. *Journal of Child Psychology and Psychiatry*, 49(5), 471-88. doi:10.1111/j.1469-7610.2007.01861.x
- World Health Organization. (2012). Depression (Fact Sheet No. 369). Retrieved from

- http://www.who.int/mediacentre/factsheets/fs369/en/
- Yeager, D. S., & Walton, G. M. (2011). Social-psychological interventions in education: They're not magic. *Review of Educational Research*, 81(2), 267-301. doi:10.3102/0034654311405999
- Yeager, D. S., Trzesniewski, K., & Dweck, C. S. (2013). An implicit theories of personality intervention reduces adolescent aggression in response to victimization and exclusion. *Child Development*, 84(3), 970-988. doi:10.1111/cdev.12003
- Yeager, D. S., Trzesniewski, K., Tirri, K., Nokelainen, P., & Dweck, C. S. (2011). Adolescents' implicit theories predict desire for vengeance: Correlational and experimental evidence. *Developmental Psychology*, 47(4), 1090-1107. doi:10.1037/a0023769
- Yeager, D.S., Johnson, R., Spitzer, B., Trzesniewski, K., Powers, J., & Dweck, C.S. (2014). The far-reaching effects of believing people can change: Implicit theories of personality shape stress, health, and achievement during adolescence. *Journal of Personality and Social Psychology*, 106(6), 867-884. doi:10.1037/a0036335
- Young, J. E. (2006). *Young Schema Questionnaire-3*. New York, USA: Cognitive Therapy Center.